CLINICAL TRIAL: NCT05200572
Title: Feasibility of a Dyadic Life Review Intervention for Older Patients With Advanced Cancer and Mild Cognitive Impairment (MCI) and Their Caregivers
Brief Title: Study of a Behavioral Intervention for Older Advanced Cancer Patients and Their Caregivers
Acronym: DLR Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lee Kehoe, Research Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006662; T32CA102618 (NIH); P30AG064103 (NIH)
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cancer, Advanced; Cognitive Impairment, Mild
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total subjects (Experimental): We will enroll dyads (defined as a pair of two people). The dyads are made up of a patient with cancer and their caregiver. The patient and caregiver dyad will go through the Dyadic Life Review intervention together. Dyadic Life Review will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes. Both patients and caregivers will each complete their own measures before and after completing the Dyadic Life Review intervention.
  Interventions: Behavioral: Dyadic Life Review (DLR)

INTERVENTIONS:
Behavioral: Dyadic Life Review (DLR) — DLR will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes. Each session will facilitate a recall of each phase of life: childhood, adolescence, young adulthood, mid-life, earlier later life, and later life. While together, the patient and caregiver will each be asked structured questions to prompt reminiscence of memories from that phase of life.

SUMMARY:
The purpose of this study is to test the feasibility of a telehealth Dyadic Life Review (DLR), adapted from individual Life Review Therapy, with patients and caregivers of older adults with advanced cancer, including those with also Mild Cognitive Impairment (MCI). The study will enroll aim to enroll 20 dyads (pairs) of patients and caregivers (40 total subjects).

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥ 65
* Able to provide informed consent. All patients will be assessed using the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) 56 - a score >14.5 will define ability to independently provide informed consent.
* Eligible patients have Stage III or IV cancer of any type
* Additionally, at least 20 patients will have a will have a high likelihood of MCI based on screening score of <26 on the Montreal Cognitive Assessment (MoCA) within their eRecord chart.
* Able to read and understand English

Patient Exclusion Criteria:

* Patients scoring <14.5 on the UBACC
* Unable to identify caregiver to participate in study

Caregiver Inclusion Criteria:

* One caregiver for each patient will be eligible and must be chosen by the patient. For the purposes of this study, a caregiver is defined as a valued and trusted person in a patient's life who is supportive in health care matters by providing valuable social support and/or direct assistive care.
* Caregivers will be selected by the patient when asked if there is a "family member, partner, friend or caregiver with whom you discuss or who can be helpful in health-related matters;" patients who cannot identify such a person ("caregiver") will remain eligible for the study.
* Age 50 or older
* Ability to provide consent
* Proficient in English

Caregiver Exclusion Criteria

* Caregivers unable to understand the consent form due to cognitive, health or sensory impairment will be excluded

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 patients were approached for consent.
Pre-assignment Details: We approached 42 patients for consent. We enrolled 38 individual patients in the DLR Intervention study.
Groups:
- DLR Intervention: Dyadic Life Review will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes.
  Dyadic Life Review (DLR): DLR will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes. Each session will facilitate a recall of each phase of life: childhood, adolescence, young adulthood, mid-life, earlier later life, and later life. While together, the patient and caregiver will each be asked structured questions to prompt reminiscence of memories from that phase of life.
Period: Overall Study
Arm/Group | DLR Intervention
Started | 38
Completed | 24
Not Completed | 14
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Population: Baseline data include both patients and caregivers (total N=38). Characteristics were not separated by participant role.
Groups:
- Dyadic Life Review Intervention (Patients and Caregivers): Dyadic Life Review will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes.
  Dyadic Life Review (DLR): Dyadic Life Review (DLR) was delivered to both members of each patient-caregiver dyad. Each dyad completed 8 video sessions facilitated by a licensed clinician. DLR will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes. Each session will facilitate a recall of each phase of life: childhood, adolescence, young adulthood, mid-life, earlier later life, and later life. While together, the patient and caregiver will each be asked structured questions to prompt reminiscence of memories from that phase of life.
Arm/Group | Dyadic Life Review Intervention (Patients and Caregivers)
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Dyads That Complete the Study
Description: The number of participants that complete the entire study procedures out of the number of participants enrolled in the study. The study consisted of one patient and one caregiver (defined as a dyad) that completed the study procedures together), therefore there were 19 dyads enrolled in the study or 38 participants. The proportion of participants that completed the study was determined out of the 19 dyads enrolled.
Time Frame: week 14
Measure: Number; unit: Dyads
Groups:
- Cancer Patients: Dyadic Life Review will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes.
  Dyadic Life Review (DLR): DLR will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes. Each session will facilitate a recall of each phase of life: childhood, adolescence, young adulthood, mid-life, earlier later life, and later life. While together, the patient and caregiver will each be asked structured questions to prompt reminiscence of memories from that phase of life.
Arm/Group | Cancer Patients
Number analyzed (Participants) | 19
Dyads | 12

2. Primary Outcome: Proportion of Participants That Consent Who Are Approached for the Study
Description: The number of participants who consented for the study out of the number of eligible participants who were approached and asked if they would like to be in the study. This outcome measures the proportion of potential participants approached who provided informed consent to participate in the Dyadic Life Review (DLR) study. A total of 42 patients were approached, and 38 provided informed consent to participate.The proportion was calculated as the number who consented divided by the total number approached (38 ÷ 42 × 100 = 90.5 percent).
Time Frame: Baseline
Population: Includes all participants approached for study enrollment (N=38).
Measure: Count of Participants; unit: Participants
Arm/Group | DLR Intervention
Number analyzed (Participants) | 42
Participants | 38

3. Primary Outcome: Number of Participants Who State the Intervention is Acceptable During a Qualitative Interview
Description: The proportion of participants who completed the full study intervention and indicated that the intervention was acceptable during post-intervention qualitative interviews. Acceptability was assessed only among participants who completed all study sessions.
Time Frame: week 14
Population: Includes all participants who completed the intervention and participated in the qualitative interview. Only 12 out of 38 participants completed the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
Participants | 12

4. Secondary Outcome: Mean Change in the UCLA Loneliness Score for Caregivers
Description: UCLA Loneliness Scale assesses perceived loneliness on a 0-10 scale, with higher scores indicating greater loneliness. Mean change was calculated as week 14 score minus baseline score for caregivers who completed the measure.
Time Frame: baseline to week 14
Population: Includes 12 caregivers who completed both baseline and week 14 assessments. Data from patient participants were not collected for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | 0.64 (4.97)

5. Secondary Outcome: Mean Change in Unidimensional Relationship Closeness Scale for Caregivers
Description: This measures the quality of the relationship with the care-receiver: assesses quality of relationship between participant and family member and has demonstrated valid scores across several relationship types, including spouses and other family members. The scale of this instrument ranges from 1 to 7 with higher scores indicating more closeness. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: Caregivers who completed both assessments (N=12). Patients were not assessed for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | -0.05 (0.7)

6. Secondary Outcome: Mean Change in Perceived Stress Scale for Caregivers
Description: Measures perceived stress, scale 0-40, higher scores indicate greater stress. Mean change calculated as week 14 minus baseline for caregivers who completed the measure.
Time Frame: baseline to week 14
Population: Caregivers who completed both assessments (N=12). Patients were not assessed for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | -0.17 (2.08)

7. Secondary Outcome: Mean Change in Caregiver Reaction Scale for Caregivers
Description: Items assess both positive and negative aspects of caregiving. Subscales: role captivity, overload, relational deprivation, competence, personal gain, family beliefs, family conflict, job conflict. The scale ranges from 0 to 24 with higher scores indicating a more negative caregiver experience. Preliminary evidence for the validity and reliability of the Caregiver Reaction Scale. Mean change calculated as week 14 minus baseline for caregivers who completed the measure.
Time Frame: baseline to week 14
Population: Caregivers who completed both assessments (N=12). Data from patients were not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | -0.42 (2.07)

8. Secondary Outcome: Mean Change in Geriatric Depression Scale for Caregivers
Description: The purpose of this scale is to identify the clinical threshold of depression in older adults. The scale ranges from 0 to 15 with higher scores indicating worse depression. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated. Mean change calculated as week 14 minus baseline for caregivers who completed the measure.
Time Frame: baseline to week 14
Population: Caregivers who completed both assessments (N=12). Patients were not assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | 1.33 (2.53)

9. Secondary Outcome: Mean Change in Distress Thermometer and Problem List for Caregivers
Description: This tool is a 10-point self-report measure to capture distress and identify a list of sources of that distress. The scale ranges from 0-10 with higher scores indicating more distress. Mean change calculated as week 14 minus baseline for caregivers who completed the measure.
Time Frame: baseline to week 14
Population: Caregivers who completed both assessments (N=12). Patients were not assessed for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | -0.42 (2.43)

10. Secondary Outcome: Mean Change in Dyadic Adjustment Scale-7 for Caregivers
Description: This is a 7-item measure to assess relationship quality that ranges from 0-36 with higher scores indicating positive relationship quality. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: Caregivers who completed both assessments (N=12). Patients were not assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | 1.17 (3.93)

11. Secondary Outcome: Mean Change in Dyadic Support Questionnaire For Caregivers
Description: 18-item measure assessing perceived received and provided support. Scale 0-145, higher scores indicate better dyadic coping. Mean change calculated as week 14 minus baseline for caregivers who completed the measure.
Time Frame: baseline to week 14
Population: Overall Number of Participants Analyzed (N=12) reflects caregiver participants only; data were not collected from patient participants for this outcome.
Measure: Mean (Standard Deviation); unit: change in score pre to post intervention
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
change in score pre to post intervention | 1.83 (6.56)

12. Secondary Outcome: Mean Change in the Correlation Between Patient and Caregiver Distress
Description: Distress measured using Distress Thermometer (0-10, higher = more distress). Pearson correlation coefficient between patient and caregiver distress scores calculated at baseline and week 14; mean change = week 14 minus baseline.
Time Frame: baseline to week 14
Population: 11 patient-caregiver dyads with complete data (N=22 participants). We analyzed 11 patient distress scores and 11 caregiver distress scores to determine the mean change in the correlation between the patient and caregiver distress scores. One subject did not complete the distress score of the 12 patient and caregiver dyads (24 total subjects) who completed the study, so we analyzed the 11 patients and 11 caregivers (22 subjects) for this outcome.
Measure: Mean (Standard Deviation); unit: change in correlation coefficient (r)
Arm/Group | DLR Intervention
Number analyzed (Participants) | 22
change in correlation coefficient (r) | -0.64 (0.05)

13. Secondary Outcome: Mean Change in PROMIS29 Depression Domain For Caregivers
Description: Patient-Reported Outcomes Measurement Information System 29-item profile (PROMIS29) - Depression Domain. Scores range from 0-10, with higher scores indicating worse depression. Mean change was calculated as week 14 minus baseline. Mean change calculated as week 14 minus baseline for caregivers who completed both assessments.
Time Frame: baseline to week 14
Population: Caregivers who completed both baseline and week 14 assessments (N=12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | -3.23 (6.93)

14. Secondary Outcome: Mean Change in PROMIS29 Anxiety Domain For Caregivers
Description: PROMIS29 - Anxiety Domain. Scores range from 0-10, with higher scores indicating worse anxiety. Mean change calculated as week 14 minus baseline. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: Caregivers who completed both baseline and week 14 assessments (N=12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | 1.61 (8.31)

15. Secondary Outcome: Mean Change in PROMIS29 Physical Function Domain For Caregivers
Description: PROMIS29 - Physical Function Domain. Scores range from 0-10, with higher scores indicating worse physical function. Mean change calculated as week 14 minus baseline. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: Caregivers who completed both baseline and week 14 assessments for this domain (N=11). Participants with missing or incomplete data for this domain were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 11
score on a scale | -0.56 (1.73)

16. Secondary Outcome: Mean Change in PROMIS29 Pain Interference Domain For Caregivers
Description: PROMIS29 - Pain Interference Domain. Scores range from 0-10, with higher scores indicating more pain interference. Mean change calculated as week 14 minus baseline. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 11
score on a scale | -2.45 (7.66)

17. Secondary Outcome: Mean Change in PROMIS29 Fatigue Domain For Caregivers
Description: PROMIS29 - Fatigue Domain. Scores range from 0-10, with higher scores indicating worse fatigue. Mean change calculated as week 14 minus baseline. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: Caregivers who completed both baseline and week 14 assessments (N=12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 12
score on a scale | -1.59 (7.82)

18. Secondary Outcome: Mean Change in PROMIS29 Sleep Disturbance Domain For Caregivers
Description: PROMIS29 - Sleep Disturbance Domain. Scores range from 0-10, with higher scores indicating worse sleep disturbance. Mean change calculated as week 14 minus baseline. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 11
score on a scale | 0.28 (10.55)

19. Secondary Outcome: Mean Change in PROMIS29 Ability to Participate in Social Roles Domain For Caregivers
Description: PROMIS29 - Ability to Participate in Social Roles Domain. Scores range from 0-10, with higher scores indicating worse social role participation. Mean change calculated as week 14 minus baseline. The change in score pre and post intervention was determined by subtracting the post intervention score from the pre intervention score and the mean of the change scores was calculated.
Time Frame: baseline to week 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLR Intervention
Number analyzed (Participants) | 11
score on a scale | -0.57 (5.37)

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Groups:
- Cancer Patients and Caregivers (Dyadic Life Review Group): The Dyadic Life Review (DLR) intervention included cancer patients and their identified caregivers. Each dyad participated in 8 weekly 60-minute sessions via video conference, facilitated by a licensed clinician. Dyadic Life Review (DLR): DLR will consist of 8 sessions delivered by a trained licensed clinician (i.e, the PI or other trained clinician) via video-conferencing in weekly sessions of 60 minutes. Each session will facilitate a recall of each phase of life: childhood, adolescence, young adulthood, mid-life, earlier later life, and later life. While together, the patient and caregiver will each be asked structured questions to prompt reminiscence of memories from that phase of life.
Arm/Group | Cancer Patients and Caregivers (Dyadic Life Review Group)
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT05200572/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT05200572/ICF_001.pdf